CLINICAL TRIAL: NCT00719147
Title: Avascular Necrosis of Weight-Bearing Joints In Patients With Hematologic Malignancies Treated With Dexamethasone Or Prednisone
Brief Title: AVN of Weight-Bearing Joints In Patients With Hematologic Malignancies Treated With Dexamethasone Or Prednisone
Status: Completed | Type: Observational
Sponsor: St. Jude Children's Research Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: AVN2
Record Dates: First submitted 2008-07-17; First posted 2008-07-21 (Estimated); Last update posted 2011-09-27 (Estimated); Status verified 2011-09

CONDITIONS: Avascular Necrosis; Acute Lymphoblastic Leukemia
MeSH Terms: conditions — Osteonecrosis; Precursor Cell Lymphoblastic Leukemia-Lymphoma | interventions — Functional Status

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- 1
  Interventions: Procedure: MRI; Other: Functional Status and Symptom Questionnaire

INTERVENTIONS:
Procedure: MRI — Not performed for study purposes, MRI will be done as part of routine clinical visit. Findings will be used for study.
Other: Functional Status and Symptom Questionnaire — Questionnaire

SUMMARY:
The primary purpose of this study is to compare the incidence of AVN in children with hematologic malignancies treated with prednisone versus dexamethasone during continuation.

DETAILED DESCRIPTION:
Patients with acute lymphoblastic leukemia enrolled on the St. Jude Children's Research Hospital front-line Acuter Lymphoblastic Leukemia protocol, Total XIIIB or the front-line Non Hodgkin's Lymphoma protocol NHL13 from 11/94 to 6/98, in continuous complete remission or who have an MRI-confirmed diagnosis of AVN of the hip or knee prior to relapse are eligible for this study.

Patients will receive an MRI examination of the hips and knees based on the following:

1. Patients who have no previous diagnosis of AVN and no previous MRI of the hips and knees will have a MRI of the hips and knees after the patient completes therapy.
2. Patients who have no previous diagnosis of AVN and have had a previous MRI of the hips and knees after completion of therapy will need no further imaging. If the patient had not completed therapy at the time of the MRI, she/he will undergo MRI of hips and knees.
3. For patients with a previous AVN diagnosis and previous MRI of the hips and knees*, the first MRI which showed AVN will be used and plain radiographs of affected joints, if not already done, will be done.

   *If a previous MRI showed AVN, but plain radiographs were not performed, the patient will have MRI and plain radiographs after enrollment in AVN2. If MRI of both hips and both knees with plain radiographs of affected joints have been done previously, the patient requires no further imaging but still will be enrolled on the study for the purpose of analysis.
4. Patients who have a previous diagnosis of AVN and no previous MRI of the hips and knees will have a MRI evaluation of the hips and knees and plain radiographs of affected joints.

Patients will be referred to a bone doctor as needed.

Patients will be asked to fill out a questionnaire (which will take approximately 10 minutes) about any pain or problems that have with their hips and knees.

If patients have already agreed to take part in the PGEN4 or PGEN5 research study; studies researching how genes affect the way the body uses certain chemotherapy drugs, genetic information from the blood tests done as part of those studies will be used to see if it can be predicted who has the greatest risk of AVN.

All study tests will be done on one day.

ELIGIBILITY:
Inclusion Criteria:

* Patients with acute lymphoblastic leukemia enrolled on the SJCRH front-line ALL protocol, TOTAL XIIIB or the front-line NHL protocol NHL13 from 11/94 to 6/98.
* Patients must be in continuous complete remission or have an MRI-confirmed diagnosis of AVN of the hip or knee prior to relapse.

Exclusion Criteria:

-

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients with acute lymphoblastic leukemia enrolled on the SJCRH front-line ALL protocol, TOTAL XIIIB or the front-line NHL protocol NHL13 from 11/94 to 6/98
Sampling Method: Non-Probability Sample
Enrollment: 170 (Actual)
Dates: Start 2001-07; Primary Completion 2005-07 (Actual); Study Completion 2005-07 (Actual)

PRIMARY OUTCOMES:
To compare the incidence of AVN in children with hematologic malignancies treated with prednisone versus dexamethasone during continuation | 7-8 years

CONTACTS AND LOCATIONS:
Overall Officials: Scott Howard, MD, Principal Investigator — St. Jude Children's Research Hospital
Locations (1):
- St. Jude Children's Research Hospital, Memphis, Tennessee, United States

REFERENCES:
- See also: St. Jude Children's Research Hosiptal — http://www.stjude.org